CLINICAL TRIAL: NCT01450683
Title: A Phase 2 Study of Itraconazole in Castrate-resistant Prostate Cancer Post-chemotherapy
Brief Title: Study of Itraconazole in Castrate-resistant Prostate Cancer (CRPC) Post-chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sandy Srinivas, Associate Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-19413; SU-12032010-7271 (Other: Stanford University); PROS0037 (Other: OnCore)
Record Dates: First submitted 2011-09-30; First posted 2011-10-12 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer; Prostatic Neoplasms; Castrate-resistant Prostate Cancer (CRPC); Androgen-insensitive Prostate Cancer; Hormone-refractory Prostate Cancer; Metastatic Disease
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Itraconazole (Experimental): 600 mg/day oral (PO)
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — 600 mg/day oral (PO)
  IUPAC name: (2R,4S)-rel-1-(Butan-2-yl)-4-{4-[4-(4-{[(2R,4S)-2-(2,4-dichlorophenyl)-2-(1H-1,2,4-triazol-1-ylmethyl)-1,3-dioxolan-4-yl]methoxy}phenyl)piperazin-1-yl]phenyl}-4,5-dihydro-1H-1,2,4-triazol-5-one
  Other Names: Sporanox; R51211

SUMMARY:
This study evaluates if itraconazole causes a reduction in the serum levels of prostate-specific antigen (PSA) in male subjects with castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
Castration-resistant prostate cancer (CRPC) is also known as "androgen-insensitive" or "hormone-refractory" prostate cancer. While numerous therapies impact biochemical response in the setting of CRPC, there remains unmet medical need, largely expressed as the lack of durable response. New therapies that extend survival of patients beyond that provided by chemotherapy are needed.

It is hypothesized that the triazole antifungal drug itraconazole, through its activity as a potent inhibitor of the Hedgehog (Hh) signaling pathway via the Smoothened (Smo) pathway, may provide clinical benefit in the treatment of prostate cancer. The Hh signaling pathway is a critical embryonic developmental pathway whose aberrant activity has been implicated in the growth and metastases of a variety of tumor types including prostate cancer. Itraconazole is structurally related to ketoconazole, demonstrated to reduce serum PSA by more than 50% in about 20 to 25% of treated prostate cancer subjects.

This study will assess efficacy on the basis of serum levels of PSA, an established surrogate endpoint for efficacy in prostate cancer.

ELIGIBILITY:
INCLUSION CRITERIA

* Male aged ≥ 18 years
* Life expectancy ≥ 6 months
* Histologically- or cytologically-confirmed adenocarcinoma of the prostate
* Metastatic disease or prior history of metastases, as documented by positive bone scan or metastatic lesions on CT or MRI
* Prostate cancer progression, as documented by PSA according to PCWG2 or radiographic progression according to RECIST criteria version 1.1
* Progression must have been during or after docetaxel based chemotherapy.
* Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM). If the patient is currently being treated with LHRH agonists (patient who have not undergone an orchiectomy), this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and treatment must be continued throughout the study.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Hemoglobin ≥ 10.0 g/dL
* Platelet count ≥100,000 microliters
* Serum creatinine ≤ 2, OR a calculated creatinine clearance ≥ 40 mL/min
* Serum bilirubin < 1.5 x ULN (except for patients Gilbert's disease)
* AST or ALT < 2.5 x ULN
* Able to swallow the study drug whole as a tablet
* Willing and able to provide written informed consent

EXCLUSION CRITERIA

* Known brain metastasis
* Radiation therapy within 4 weeks of Cycle 1, Day 1
* Prior systemic treatment with an azole drug (eg, fluconazole, ketoconazole) within 4 weeks of Cycle 1, Day 1
* Prior flutamide (Eulexin) treatment within 4 weeks of Cycle 1, Day 1 (patients whose PSA did not decline for ≥ 3 months months in response to antiandrogen given as a 2nd line or later intervention will require only a 2-week washout prior to Cycle 1,Day 1)
* Prior Bicalutamide (Casodex), nilutamide (Nilandron) treatment within 6 weeks of Cycle 1 Day 1 (patients whose PSA did not decline for ≥ 3 months in response to antiandrogen given as a 2nd line or later intervention will require only a 2-week washout prior to Cycle 1 Day 1)
* Known active or symptomatic viral hepatitis or chronic liver disease
* Clinically significant heart disease as evidenced by myocardial infarction or arterial thrombotic events in the past 6 months; severe or unstable angina
* Other malignancy, except non-melanoma skin cancer, with a ≥ 30% probability of recurrence within 24 months
* Administration of an investigational therapeutic within 30 days of Cycle 1, Day 1
* Any condition which, in the opinion of the investigator, would preclude the patient's participation in this trial.
* No more than 3 prior chemotherapy regimens.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sandy Srinivas, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Itraconazole
Started | 4
Completed | 2
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Castrate-resistant Prostate Cancer Patients
Arm/Group | Itraconazole
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 78 [73 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Serum PSA
Description: Number of subjects with > 50% drop in serum PSA as compared to baseline, at 12 weeks and confirmed at 15 weeks
Time Frame: 12 weeks treatment, with primary outcome assessed at 15 weeks
Measure: Number; unit: participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 4
participants | 0

ADVERSE EVENTS:
Arm/Group | Itraconazole
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itraconazole (N=4)
Other-Nocturia (Renal and urinary disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Other-Sneezing (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Other-Decreased Hearing (Ear and labyrinth disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Facial Flushing (Vascular disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Other-Shoulder Pain (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (1)
Edema Limbs (Gastrointestinal disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No